CLINICAL TRIAL: NCT05320133
Title: The Effect and Safety of Jinghua Weikang Capsule Containing Quadruple Therapy for IgAN With Helicobacter Pylori Infection, a Randomized Pilot Study
Brief Title: Jinghua Weikang Capsule Containing Quadruple Therapy for IgAN With Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021CR36
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; IgA nephropathy; Jinghua Weikang Caplsule; Bismuth-containing quadruple therapy; Eradication
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JWC group (Experimental): Jinghua Weikang Capsule containing quadruple therapy.
  Interventions: Drug: JWC containing quadruple therapy
- Control group (Active Comparator): Bismuth-containing quadruple therapy.
  Interventions: Drug: Bismuth-containing quadruple therapy

INTERVENTIONS:
Drug: JWC containing quadruple therapy — Subjects will receive the rabeprazole 10mg, moxycillin 1.0g, clarithromycin 500mg and Jinghua Weikang Capsule 240mg twice daily for 14 days.
  Arms: JWC group
Drug: Bismuth-containing quadruple therapy — Subjects will receive the rabeprazole 10mg, moxycillin 1.0g, clarithromycin 500mg and bismuth potassium citrate 220mg twice daily for 14 days.
  Arms: Control group

SUMMARY:
This study is to evaluate the efficacy and safety of the Jinghua Weikang Capsule (a Chinese patent medicine for peptic ulcer and gastritis) containing quadruple therapy (Jinghua Weikang Caplsule plus triple therpy) for eradicating Helicobacter pylori in IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* IgA nephropathy diagnosed by renal biopsy;
* Current Helicobacter pylori infection;
* Age 18-65.

Exclusion Criteria:

* ①eGFR<90ml/（min·1.73m2）-
* History of Helicobacter pylori treatment
* Present taking hormones or immunosuppressants
* Malignant tumor and high-grade intraepithelial neoplasia and severe dysplasia of gastric mucosa
* Allergy history to medicines used in the study
* History of gastric surgery
* Uncontrolled chronic diseases such as diabetes, cardiovascular and cerebrovascular diseases, respiratory diseases, mental disorders and other researchers are considered to affect treatment and assessment
* Combined with other primary or secondary nephropathy except for IgAN
* Combined with acute renal injury
* Female patients with pregnancy, lactation and planned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradicaion rate | The forth week after the treatment.
  The Helicobacter pylori infection status was measured by 13-carbon breath test.

SECONDARY OUTCOMES:
Blood creatinine level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average blood creatinine level between two groups.
Blood urea nitrogen level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average blood urea nitrogen level between two groups.
eGFR | Baseline, the third and sixth month after the treatment, respectively.
  The change of average eGFR level between two groups.
24hrs urine protein level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average24hrs urine protein level between two groups.
Blood presure | Baseline, the third and sixth month after the treatment, respectively.
  The change of average blood presure level between two groups.
IgA level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average IgA level level between two groups.
IgA1 level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average IgA1 level between two groups.
Gd-IgA1 level | Baseline, the third and sixth month after the treatment, respectively.
  The change of average Gd-IgA1 level level between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: HUI YE, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on https://clinicaltrials.gov.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be uploaded within 6 month after Dec 31, 2024.
Access Criteria: The user of ClinicalTrials.gov PRS could access the data.

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639